CLINICAL TRIAL: NCT01683903
Title: Comparison of Cardiac Rehabilitation Benefits Between Coronary and Non-coronary Patients Through a 24 Months Follow-up : the "INCARD" Study
Brief Title: Comparison of Cardiac Rehabilitation Benefits Between Coronary and Non-coronary Patients Through a 24 Months Follow-up After Myocardial Infarction: the "INCARD" Study
Acronym: INCARD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Sud Francilien (Other)
Responsible Party: Principal Investigator, KOUKOUI Francois, MD, Centre Hospitalier Sud Francilien
Other Study IDs: INCARD
Record Dates: First submitted 2012-08-10; First posted 2012-09-12 (Estimated); Last update posted 2012-09-12 (Estimated); Status verified 2012-09

CONDITIONS: Heart Failure
Keywords: heart failure; cardiac rehabilitation; myocardial infarction
MeSH Terms: conditions — Heart Failure; Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Non coronary patients (NC): Patient with myocardial infarction with non-coronary (NC) etiology
- Coronary patients (C): Patients with myocardial infarction due to coronary disease

SUMMARY:
Treatment of chronic heart failure requires multidisciplinary approaches with a recognized role for cardiac rehabilitation. Rehabilitation helps to improve patient's functional, decrease morbidity and mortality, decrease rehospitalization rate, thereby reducing costs of this disease. After recovery from the acute phase of cardiac infarction, patients admitted to the rehabilitation center will follow the usual rehabilitation program during the hospitalization period. This step precludes outpatient follow-up period in our day hospital, in accordance with their physicians and cardiologists who manage the monitoring. The study INCARD (Insuffisance Cardiaque en Readaptation Durable) will be developed to evaluate the benefits of a sustainable rehabilitation heart failure on patients treated optimally and educated during a follow-up period of 24 months. The main objective of the study will be to compare the benefits of rehabilitation between coronary (C) and non-coronary (NC) patients for each evaluation time point, periodically recorded

DETAILED DESCRIPTION:
We will undertake a prospective follow-up study of 150 rehabilitated patients with heart failure (75 C; 75 NC). The main objective will be to compare the benefits of rehabilitation between coronary and non-coronary patients based on functional improvement i.e. improvements of VO2max, LVEF (ultrasound method and/or isotopic), 6-min walk test, Minnesota index of quality of life. In addition, clinical outcomes (HR, SBP, DBP, BMI) and paraclinical data (creatinine clearance) will be measured as patients' standard clinical follow-up .

Clinical data of the patients admitted to the cardiac rehabilitation, including heart failure patients (LVEF <40), will be recorded after collection of their signed informed consent agreement. Patients will be addressed from heart failure intensive care units for coronary (USIC) or acute cardiac services to the rehabilitation department. Patients will be admitted in the rehabilitation department when there are clinically stable (at least three weeks after the acute episode). Etiology of the heart failure will be assessed and patients stratified as C or NC patients.

Expected Results We will estimate the mean duration of inpatient rehabilitation (H period). Then, we will follow patients' cardiac evaluation parameters recorded from an outpatient follow-up, first 3 months after inclusion and then every 6 months over the 24 months of outpatient follow-up.

These data will allow for comparison of the benefits of rehabilitation between coronary (C) and non-coronary (NC) patients for each evaluation time point and will give information on the clinical improvement of each group of patients.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years old,
* Signed informed consent,
* Patients with left ventricular ejection fraction below 40 %,
* Stable for over 3 weeks,
* Known etiology,
* Able to do the performance test on treadmil or bicycle in order to have rehabilitation.
* No clinical avoidance reasons.
* Patient with health care registration.
* Agreement from the general practictioner and from the cardiologist that follows the patient.

Exclusion Criteria:

* Age below 18 years old,
* Unstable heart failure,
* Unable to do a performance test as indicated above,
* Patients not able to understand clinical counseling.
* Patient under tutella.
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic heart failure patients
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2012-08; Primary Completion 2014-08 (Estimated); Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
Change in VO2max every 6 months over the 24 months | every 6 months over the 24 months of outpatient follow-up
  VO2max (L)
Change in Left ventricular ejection fraction every 6 months over the 24 months of outpatient follow-up | every 6 months over the 24 months of outpatient follow-up
  Left ventricular ejection fraction (ultrasound method and/or isotopic) in %
Change on 6-min walk test every 6 months over the 24 months | every 6 months over the 24 months of outpatient follow-up
  6-min walk test (m)
Change on Minnesota index of quality of life every 6 months over the 24 months | every 6 months over the 24 months of outpatient follow-up
  Minnesota index of quality of life.
Change on heart rate every 6 months over the 24 months | every 6 months over the 24 months of outpatient follow-up
  Heart rate (bpm)
Change on systolic blood pressure every 6 months over the 24 months | every 6 months over the 24 months of outpatient follow-up
  systolic blood pressure (mmHg)
Change on diastolic blood pressure every 6 months over the 24 months | every 6 months over the 24 months of outpatient follow-up
  diastolic blood pressure (mmHg)
Change on body mass index every 6 months over the 24 months | every 6 months over the 24 months of outpatient follow-up
  Measurement of weight and height, calculation of body mass index (kg/m2)
Change on creatine clearance every 6 months over the 24 months | every 6 months over the 24 months of outpatient follow-up
  creatine clearance (ml/min)

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalien Sud Francilien, Corbeil, France

REFERENCES:
- [Background] Dickstein K, Cohen-Solal A, Filippatos G, McMurray JJ, Ponikowski P, Poole-Wilson PA, Stromberg A, van Veldhuisen DJ, Atar D, Hoes AW, Keren A, Mebazaa A, Nieminen M, Priori SG, Swedberg K; ESC Committee for Practice Guidelines (CPG). ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure 2008: the Task Force for the Diagnosis and Treatment of Acute and Chronic Heart Failure 2008 of the European Society of Cardiology. Developed in collaboration with the Heart Failure Association of the ESC (HFA) and endorsed by the European Society of Intensive Care Medicine (ESICM). Eur Heart J. 2008 Oct;29(19):2388-442. doi: 10.1093/eurheartj/ehn309. Epub 2008 Sep 17. No abstract available. PMID 18799522
- [Derived] Koukoui F, Desmoulin F, Lairy G, Bleinc D, Boursiquot L, Galinier M, Smih F, Rouet P. Benefits of cardiac rehabilitation in heart failure patients according to etiology: INCARD French study. Medicine (Baltimore). 2015 Feb;94(7):e544. doi: 10.1097/MD.0000000000000544. PMID 25700319